CLINICAL TRIAL: NCT01781624
Title: Evaluation of an Oral Nutritional Supplement With a New Protein Blend
Brief Title: Evaluation of an Oral Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BL13
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Gastro-intestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Oral Nutritional Supplement (Experimental): 2 containers a day of a high calorie, complete, balanced, ready-to-drink oral nutritional supplement with a new protein blend.
  Interventions: Other: Study Oral Nutritional Supplement

INTERVENTIONS:
Other: Study Oral Nutritional Supplement — Supplement contains a new protein mix consisting of a blend of milk, soy, and pea protein.

SUMMARY:
The objective of this study is to evaluate gastrointestinal tolerance of an oral nutritional supplement containing a new protein blend in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the study if they meet all of the following inclusion criteria:

1. Age ≥ 60 and ≤ 90 years
2. Body Mass Index (BMI) > 20 but < 35

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. History of diabetes
2. Currently taking or has taken antibiotic within 1 week prior to enrollment
3. Major surgery less than 3 months prior to enrollment in the study
4. Current active malignant disease or was treated within the last 6 months for cancer
5. Immunodeficiency disorder
6. Myocardial infarction within the last 3 months prior to enrollment
7. Chronic obstructive pulmonary disease (COPD)
8. Allergy to any of the ingredients in the study product
9. Aversion to flavor of product being tested
10. Obstruction of the gastrointestinal tract precluding ingestion or absorption of the study product, inflammatory bowel disease, ulcer, gastric reflux disease, short bowel syndrome, or other major gastrointestinal disease
11. Dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder
12. Pursuing or has unintentional weight loss or weight gain ≥ 5% in last 4 weeks
13. Medications/dietary supplements/substances that could profoundly modulate metabolism or affect GI motility

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Study Day 1-7
  Self-reported questionnaire

SECONDARY OUTCOMES:
Study Product Compliance | Study Day 1-7
  Self-reported number of containers consumed per day
Weight | Study Day 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Nelson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Radiant Research, Inc., Cincinnati, Ohio, United States